CLINICAL TRIAL: NCT05846958
Title: Efficacy of Laser Acupuncture on Neurophysiological Parameters of Median Nerve in Postpartum Women: A Randomized Controlled Clinical Trial
Brief Title: Efficacy of Laser Acupuncture on Neurophysiological Parameters of Median Nerve in Postpartum Women
Acronym: CTSLA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Afaf Mohamed Botla, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Postpartum CTS
Record Dates: First submitted 2023-04-06; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Neurophysiologic Abnormality

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser acupuncture (Experimental): Each patient in this group will receive laser acupuncture based on the recommended LLLT treatment doses for CTS of the World Association of Laser Therapy.
  Interventions: Device: laser acupuncture; Device: night splint
- control group (Active Comparator): Each patient in this group will wear night splint every night for 4 weeks
  Interventions: Device: night splint

INTERVENTIONS:
Device: laser acupuncture — Each patient in experimental group will receive laser acupuncture for 10 s with at least 4J/point for each point.10 minutes, three times per week for 4 weeks (total of 12 sessions)
  nieght splint for 4 weeks .
  Arms: laser acupuncture
Device: night splint — wearing night splint for 4 weeks

SUMMARY:
BACKGROUND: Carpal tunnel syndrome (CTS), the most common entrapment neuropathy of the upper extremity, is caused by compression of the median nerve as it travels through the carpal tunnel CTs is a very common complication found in pregnancy, which is reported as high as 62% in pregnant females. The functioning of median nerve is compromised in almost all pregnant females especially during the third trimester of pregnancy, the majority may still feel some symptoms up to 3 years after delivery. Many clinicians have used LLLT on acupuncture points, which is called laser acupuncture (LA), to treat many clinical problems, such as musculoskeletal pain, lateral epicondylitis, headaches, etc. In contrast with traditional acupuncture needles, LA is a non-invasive therapy that does not cause tingling/pain during procedures Objective: to determine efficacy of laser acupuncture on electrophysiological parameters of median nerve in postpartum women

DETAILED DESCRIPTION:
Intervention description

1. Experimental Group:

   Each patient in this group will receive laser acupuncture on PC4 (Ximen), PC6 (Neiguan), PC7 (Daling), PC8 (Laogong), LI4 (Hegu), LI10 (Shousanli), LI11 (Quchi), HT3 (Shaohai), HT7 (Shenmen), LU10 (Yuji) acupoints in addition to wearing night splint. LA will be applied to each acupuncture point for 10 s with at least 4J/points based on the recommended LLLT treatment doses for CTS of the World Association of Laser Therapy.
2. Control Group:

Each patient in this group will wear night splint every night for 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* Their BMI will be range from 25 to 30 Kg/m2.
* The electrophysiological evidence of mild or moderate median nerve lesion at wrist (mild: sensory nerve latency >3.5 ms at third digit, moderate: sensory nerve latency >3.5 ms at third digit and median motor latency>4.2 ms)
* Positive phalen's test.
* Positive tinel's test.
* Carpal tunnel of dominant hand could be participated.

Exclusion Criteria:

* History of brachial plexopathy or malignancy.
* Radial, ulnar neuropathy, proximal median neuropathy or polyneuropathy.
* Previous wrist surgery or steroid injection for carpal tunnel syndrome.
* History of trauma, fracture, deformity or inflammation in the wrist, such as rheumatoid arthritis.
* Coagulation abnormalities, pregnancy, fever and infections.
* Skin disease and skin cancer.
* Spots, birthmarks or tattoos over the work points. 8- Pacemaker and implementable medical devices.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Postpartum women with mild to moderate carpal tunnel syndrome will participate in this study
Enrollment: 50 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-20 (Estimated); Study Completion 2023-07-28 (Estimated)

PRIMARY OUTCOMES:
sensory nerve conduction velocity (SNCV) measured in m/s | 4 weeks
  will be measured at the beginning of the study and at the end of the treatment program througth EMG

SECONDARY OUTCOMES:
Hand grip strength in Kg | 4 weeks
  will be measured at the beginning of the study and at the end of the treatment program using pinch grip dynamometer
Symptoms severity and functional capacity (Score) | 4 weeks
  will be measured at the beginning of the study and at the end of the treatment program using Boston symptoms severity scale (BSSS)

CONTACTS AND LOCATIONS:
Overall Officials: Afaf M Botla, Professor, Principal Investigator — Cairo University
Locations (1):
- Out clinic, Faculty of physical therapy, Dokki, Giza Governorate, Egypt